CLINICAL TRIAL: NCT05137847
Title: Post-marketing Observational Study of Remitoro® Intravenous Injection 300 μg - Safety of Remitoro in Patients With Recurrent or Refractory Peripheral T Cell Lymphoma and Cutaneous T Cell Lymphoma (All Case Study)
Brief Title: A Study of Remitoro in Participants With Recurrent or Refractory Peripheral T Cell Lymphoma and Cutaneous T Cell Lymphoma (All Case Study)
Status: Completed | Type: Observational
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E7777-M081-501
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Lymphoma, T-cell, Peripheral; Lymphoma, T-cell, Cutaneous
Keywords: Peripheral T cell lymphoma; Cutaneous T cell lymphoma; Remitoro; E7777; Adverse drug reactions
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous; Drug-Related Side Effects and Adverse Reactions | interventions — denileukin diftitox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Remitoro: Participants with recurrent or refractory peripheral T cell lymphoma (PTCL) and cutaneous T cell lymphoma (CTCL) will be administered with Remitoro 9 microgram per kilogram (mcg/kg), intravenous (IV) infusion, over 1 hour once daily for 5 consecutive days followed by 16 days withdrawal period in a 21 day cycle (up to maximum of 8 cycles). The dosage will be adjusted depending on the condition of the participant. All the participants will be observed for up to 24 weeks prospectively.
  Interventions: Drug: Remitoro

INTERVENTIONS:
Drug: Remitoro — Intravenous infusion.
  Other Names: Denileukin diftitox

SUMMARY:
The primary purpose of the study is to investigate the incidence of adverse drug reactions (ADRs) (ADR of special interest: capillary leak syndrome, infusion reaction, rhabdomyolysis, myelosuppression, infection, hepatic dysfunction, visual impairment/color blindness, ischemic heart disease/arrhythmia/cardiac failure, and severe skin disorders).

ELIGIBILITY:
Inclusion Criteria:

1. Participants with PTCL or CTCL.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with recurrent or refractory PTCL or CTCL administered Remitoro will be included in this study.
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with ADR | Up to Week 24
  Incidence of ADR, especially for capillary leak syndrome, infusion reaction, rhabdomyolysis, myelosuppression, infection, hepatic dysfunction, visual impairment/color blindness, ischemic heart disease/arrhythmia/cardiac failure, and severe skin disorders will be assessed. An ADR is defined as harmful and unintended responses to the normal administration/use of drugs, in which a causal relationship with the drug in question cannot be ruled.

SECONDARY OUTCOMES:
Percentage of Participants With Best Overall Response (BOR) | Up to Week 24
  Percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on physician assessment will be determined. PTCL is evaluated according to revised response criteria for malignant lymphoma (Cheson, 2007). CTCL is evaluated according to clinical endpoints and response criteria in mycosis fungoides and sezary syndrome (Olsen, 2011). CR: Disappearance of all evidence of disease; PR: Regression of measurable disease and no new sites.

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Eisai Trial Site 3, Nagoya
  - Eisai Trial Site 1, Osaka
  - Eisai Trial Site 2, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.